CLINICAL TRIAL: NCT00714818
Title: Genetic Counseling for Female First Degree Relatives of Individuals With Mental Illness: Impact on Knowledge, Risk Perception, Perceived Control and Internalized Stigma.
Brief Title: Impact of Genetic Counseling for Female First Degree Relatives of Individuals With Mental Illness
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: H07-02706
Record Dates: First submitted 2008-07-08; First posted 2008-07-14 (Estimated); Last update posted 2011-11-23 (Estimated); Status verified 2011-11

CONDITIONS: Schizophrenia; Bipolar Disorder; Schizoaffective Disorder
Keywords: Schizophrenia; Bipolar Disorder; Schizoaffective disorder; Genetic Counseling; Risk perception; Stigma; Control; Knowledge; family members; Sibling parent or child with schizophrenia; Sibling parent or child with bipolar disorder; Sibling parent or child with schizoaffective disorder
MeSH Terms: conditions — Schizophrenia; Bipolar Disorder; Psychotic Disorders; Social Stigma | interventions — Genetic Counseling

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- GC (Experimental): One face-to-face genetic counseling session of 1-2hours duration, with a board certified or board eligible genetic counselor which will involve, documentation of a detailed family history, discussion of: the contributors to mental illness pathogenesis, illness risk reduction strategies, chances for family members to develop mental illness (if required), supportive counseling around living with illness/risk of illness/managing illness vulnerability, and referral to support organizations as required.
  Interventions: Behavioral: Genetic Counseling
- EB (Active Comparator): Educational Booklet: One educational booklet that provides information about the causes of mental illnesses, and the chances for relatives of affected individuals to develop mental illness will be provided to participants
  Interventions: Behavioral: Genetic Counseling
- WT (No Intervention): Waitlist

INTERVENTIONS:
Behavioral: Genetic Counseling — One face-to-face genetic counseling session of 1-2hours duration, with a board certified or board eligible genetic counselor which will involve, documentation of a detailed family history, discussion of: the contributors to mental illness pathogenesis, illness risk reduction strategies, chances for family members to develop mental illness (if required), supportive counseling around living with illness/risk of illness/managing illness vulnerability, and referral to support organizations as required
  Arms: GC
Behavioral: Genetic Counseling — One educational booklet that provides information about the causes of mental illnesses, and the chances for relatives of affected individuals to develop mental illness will be provided to participants.
  Arms: EB

SUMMARY:
Women with a close relative who has experienced mental illnesses like schizophrenia, bipolar disorder or schizoaffective disorder often have a poor understanding of the causes of the illness, and are often very worried about the chance that any children that they have will become affected with the same illness. Often, because of this fear, these healthy women choose not to have children.

Genetic counseling is a process where information about the causes of illnesses, and about chances for family members of individuals with these illnesses to become similarly affected is provided in a supportive environment by a specially trained healthcare professional. This study will investigate whether genetic counseling can reduce perceptions of risk and stigma, and increase perceived control and knowledge about the causes of the illness, amongst women who have a first degree relative with a major mental illness.

DETAILED DESCRIPTION:
We will recruit 75 women who have a close relative with a major psychiatric disorder (as defined above). Each participant will be randomized into one of 3 groups of approximately equal size: one of which will receive genetic counseling within 1 month after enrollment (GC), another will receive the educational brochure within 1 month (EB), and the last will be assigned to waitlist (WT). After randomization (but prior to intervention for GC and EB groups, and within 1 month after enrollment for the WT group) we will gather baseline information regarding the 4 outcome measures (perceived risk and control, stigma, and knowledge). We will re-assess the 4 outcome measures immediately post-intervention for GC and EB groups. A further follow-up (for all groups) will be conducted two months after enrollment (which is 1 month post intervention for GC and EB groups).

ELIGIBILITY:
Inclusion Criteria:

* Fluent in English, and
* Have a first degree relative diagnosed with schizophrenia, bipolar, or schizoaffective disorder, and
* Reside in BC, and be able to attend 3 study visits over 1.5 months

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2008-08; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
knowledge | immediately post intervention and 1 month post intervention
risk perception | immediately post intervention and 1 month post intervention
stigma | immediately post intervention and 1 month post intervention
perceived control | immediately post intervention and 1 month post intervention

CONTACTS AND LOCATIONS:
Overall Officials: Jehannine Austin, PhD, CCGC, CGC, Principal Investigator — University of British Columbia; Catriona Hippman, Study Director — University of British Columbia; Erin Michalak, Study Director — University of British Columbia; William Honer, MD, Study Director — University of British Columbia
Locations (1):
- Centre for Complex Disorders, BC Mental Health and Addictions Reserach Institute, Vancouver, British Columbia, Canada